CLINICAL TRIAL: NCT07368179
Title: Emergency Front-of-neck Access in Infants: A Crossover Trial Evaluating Surgical and Percutaneous eFONA Techniques in a Simulated Rabbit Model
Brief Title: Neck Rescue Access Comparison
Acronym: eFONA
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Gaslini Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: FONA Riva2026
Record Dates: First submitted 2026-01-05; First posted 2026-01-26 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Tracheostomy Complication; Emergency Front of Neck Airway in Children; Anesthesia
Keywords: pediatric airway; tracheotomy; eFONA; CICO

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Percutaneous Seldinger-Guided Tracheal Access (Melker) (Active Comparator): Melker technique described in Interventions
  Interventions: Procedure: Percutaneous Seldinger-Guided Tracheal Access (Melker)
- scalpel-bougie tracheostomy (SBT) (Active Comparator): SBT Technique described in Interventions
  Interventions: Procedure: scalpel-bougie tracheostomy

INTERVENTIONS:
Procedure: Percutaneous Seldinger-Guided Tracheal Access (Melker) — 1. The operator palpates and stabilizes the trachea in the midline. A syringe is attached to the introducer needle.
  2. The needle is advanced through the skin in the midline with continuous aspiration until intratracheal placement is confirmed by free air aspiration.
  3. A flexible guidewire is inserted through the needle into the tracheal lumen.
  4. The needle is removed while maintaining the guidewire in position.
  5. A dilator with integrated airway catheter is advanced over the guidewire using controlled rotational pressure.
  6. After intratracheal placement, the dilator and guidewire are removed.
  7. The cuffed airway catheter (inner diameter 3.5 mm) is connected to a ventilation device to establish ventilation.
  Other Names: Melker
  Arms: Percutaneous Seldinger-Guided Tracheal Access (Melker)
Procedure: scalpel-bougie tracheostomy — 1. The assistant places themselves with two preparation clamps at the head end of the table and assists with each hand placed lateral to the neck, so that the operating field is freely accessible. After the trachea or cricoid is palpated, a long median longitudinal skin incision of 2-3 cm is made from the cricoid caudally 2. The assistant uses straight clamps to pull the two edges of the skin incision apart dorso-laterally. In the event of major bleeding this maneuver should allow the blood to drain off dorsally and the view of the anatomical structures should be less impaired. 3. Layer by layer of the anatomical structures are cut through with the scalpel and tightened with the clamps accordingly. 4. Using a longitudinal incision, two to three tracheal rings are cut through distally to the cricoid 5. An 8 FR Frova catheter is inserted through the orifice into trachea. 6. A tracheal tube (ID 3.0 mm) is inserted over the Frova catheter to secure the airway permanently.
  Other Names: SBT
  Arms: scalpel-bougie tracheostomy (SBT)

SUMMARY:
Emergency front-of-neck access (eFONA) represents the final lifesaving intervention in a pediatric "can't intubate, can't oxygenate" scenario. Despite its importance, there is no consensus on the optimal eFONA technique in infants, and existing evidence is limited by low-fidelity models and a lack of randomized crossover comparisons. The objective of this randomized crossover simulation trial is to compare a surgical scalpel-bougie tracheostomy technique with a percutaneous Seldinger-guided technique under standardized, high-fidelity simulated infant emergency conditions. Using a rabbit cadaver model with simulated bleeding, physiological deterioration, and anatomical constraints, the study aims to assess time to successful ventilation and procedure-related injury patterns for both techniques.

DETAILED DESCRIPTION:
With approval from the competent ethics committee, this single-center randomized crossover simulation trial will recruit board-certified pediatric anesthesiologists and pediatric intensivists. Participants will be randomized to perform either a percutaneous Seldinger-guided front-of-neck access technique or a surgical scalpel-bougie tracheostomy technique first, followed by crossover to the alternative technique.

Prior to assessment, participants will receive standardized video-based instruction for the assigned technique and will complete four supervised practice attempts on rabbit cadavers. A fifth attempt will be formally assessed. The same process will then be repeated after crossover to the second technique. Participants will be allowed to re-watch the instructional videos throughout the study.

All procedures will be performed on prepared rabbit cadavers in a high-fidelity simulated infant emergency environment. Anatomical realism will be enhanced using an infant mannequin head, shoulder roll, and standardized positioning. Psychological stress will be simulated using an audible oxygen saturation monitor with progressive desaturation and bradycardia. Physiological realism will be further enhanced by continuous simulated bleeding during the procedure using an infusion system delivering artificial blood near the trachea.

Performance time will be measured from skin contact to confirmed ventilation, defined by visible lung expansion. A procedure duration exceeding three minutes will be classified as failure. Procedure-related injuries, including damage to tracheal structures and posterior wall perforation, will be systematically documented. Each participant acts as their own control, minimizing inter-individual variability.

The study is designed to provide comparative data on performance efficiency and safety profiles of two fundamentally different pediatric eFONA techniques under realistic emergency conditions.

ELIGIBILITY:
Inclusion Criteria:

* board certified pediatric anesthesiologists or pediatric intensive care doctor
* informed consent signed

Exclusion Criteria:

* none

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02-02 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Performance Time | During the procedure; measured from initial palpation of the trachea until establishment of a secured airway with confirmed lung ventilation
  Performance time between the percutaneous Seldinger-guided tracheal access and the scalpel-bougie tracheostomy technique. If tracheal access was not achieved within two minutes, the attempt was terminated and recorded as unsuccessful.

SECONDARY OUTCOMES:
Success rate of emergency front-of-neck airway establishment | During the procedure
  Success was defined as establishment of a secured airway with confirmed lung ventilation using the assigned technique within two minutes. Confirmed lung ventilation was assessed by visible chest rise and ventilation of the lung.
  Failure was defined as inability to establish a secured airway within two minutes, leading to termination of the attempt.
rate of thyroid cartilage injuries | Immediately after the procedure (post-procedural inspection)
  Thyroid cartilage injury was assessed after each attempt by post-procedural inspection of the laryngeal framework. Injury was defined as any visible damage to the thyroid cartilage attributable to the procedure (e.g., fracture, laceration, perforation, or gross deformation). Injuries were recorded as present/absent; if present, the type of injury was documented.
rate of cricoid injuries | Immediately after the procedure (post-procedural inspection)
  Cricoid injury was assessed after each attempt by post-procedural inspection of the laryngeal framework. Injury was defined as any visible damage to the cricoid cartilage attributable to the procedure (e.g., fracture, laceration, perforation, or gross deformation). Injuries were recorded as present or absent; if present, the type of injury was documented.
number of tracheal ring damaged | Immediately after the procedure (post-procedural inspection)
  Tracheal ring damage was assessed after each attempt by post-procedural inspection of the trachea. Damage was defined as any visible injury to one or more tracheal rings attributable to the procedure (e.g., fracture, laceration, or perforation). Damage was recorded as present or absent; if present, the number of affected tracheal rings was documented.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsspital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No